CLINICAL TRIAL: NCT06630039
Title: Examination of the Validity and Reliability of the Short-Western Ontario Rotator Cuff Disability Index in Turkish in Patients With Rotator Cuff Injury
Brief Title: Turkish Validity and Reliability of Short-Western Ontario Rotator Cuff Disability Index
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Emel Mete, Research Assistant, Istanbul Medeniyet University
Other Study IDs: SHORTWORC
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Rotator Cuff Injuries
Keywords: roatator cuff injuries; scale validity; pain
MeSH Terms: conditions — Rotator Cuff Injuries; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with Rotator cuff injury: Patients with roatator cuff injury who are aged over 18 years
  Interventions: Other: Scale validity and reliability

INTERVENTIONS:
Other: Scale validity and reliability — The aim of this study is to adapt the Short-Western Ontario Rotator Cuff Disability Index (SHORTWORC) to Turkish society in patients with rotator cuff injury and to make its validity and reliability in Turkish. It has 7 questions. The patients will be sought to answer questionnaires during regular rehabilitation sessions.

SUMMARY:
The aim of this study is to adapt the Short-Western Ontario Rotator Cuff Disability Index (SHORTWORC) to Turkish society and to make its validity and reliability in Turkish. The Western Ontario Rotator Cuff Disability Index (WORC) developed by Kirkley et al assesses quality of life in patients with Rotator Cuff İnjury. The WORC has 21 questions. The WORC was shortened and renamed as Short-Western Ontario Rotator Cuff Disability Index (SHORTWORC). The SHORTWORC consists of 7 questions. This study will be conducted with patients with rotator cuff injuries. The patients will be sought to answer questionnaires during regular rehabilitation sessions. 35 participants will be included in the study. In order to evaluate the validity of the SHORTWORC, the Western Ontario Rotator Cuff Disability Index (WORC), which can evaluate the quality of life in patients with rotator cuff injury and has been validated in Turkish, and the The University of California-Los Angeles (UCLA) shoulder scale, which can evaluate the functionality of shoulder and has been validated in Turkish, will be used. Scales will be repeated after 15 days to assess test-retest reliability.

DETAILED DESCRIPTION:
The reliability and validity of the scale will begin with language equivalence and cultural adaptation. The scale will be translated from English to Turkish by two people who are fluent in Turkish and English. A single Turkish translation will be obtained from these two Turkish translations with a common opinion.

The scale, which has been translated into Turkish, will be translated into English by two other people who are fluent in Turkish and English. The scale translated into English will be compared with the original. In the pre-trial phase, a reassessment will be conducted with 15 participants to test the intelligibility of the scale. Based on the results of the pre-test phase, the final version of SHORTWORC will be able to be modified. The data of SHORTWORC are collecting through face-to-face when the patients came to the rehabilitation center. 35 participants will be included in the study.

In order to evaluate the validity of the SHORTWORC, the Western Ontario Rotator Cuff Disability Index (WORC), which can evaluate the quality of life in patients with rotator cuff injury and has been validated in Turkish, and the University of California-Los Angeles (UCLA) shoulder scale, which can evaluate the functionality of shoulder and has been validated in Turkish, will be used. Scales will be repeated after 15 days to assess test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 18 years of age who have been diagnosed with a rotator cuff injury,
* Patients whose native language is Turkish,
* Individuals with pain intensity > 2 according to the Visual Analog Scale,
* Individuals with a Mini Mental State Examination score of >24,

Exclusion Criteria:

* Individuals with pain and disability due to any shoulder pathology other than rotator cuff injury,
* Individuals who cannot read or write Turkish,
* Individuals with shoulder fractures, surgical interventions and other accompanying shoulder pathologies,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rotator cuff injury who are aged over 18 years
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Disability | baseline
  Disability will be assessed with the Short-Western Ontario Rotator Cuff Disability Index (SHORTWORC) in patients with rotator cuff injury. It haf 7 items. Each item is scored on a 0-to-100-mm visual analog scale, summing a total score ranging from 0 (best possible score) to 700 (worst possible score). Higher scores indicate poorer quality of life.

SECONDARY OUTCOMES:
Functionality of shoulder | baseline
  Functionality of shoulder will be assessed with the University of California-Los Angeles (UCLA) shoulder scale. It contains a total of 5 questions belonging to 5 categories: Pain (scored from 1-10), Function (scored from 1-10), range of motion (scored from 0-5), muscle strength (scored from 0-5), patient satisfaction (scored from 0-5). Each category is scored differently. Higher scores indicate better shoulder functionality.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - İstanbul Medeniyet University, Istanbul
  - Istanbul Medeniyet University, Istanbul

IPD SHARING:
Plan to Share IPD: No